CLINICAL TRIAL: NCT02973490
Title: Transanal Tube Drainage in Endoscopic Submucosal Dissection of the Colorectal Tumor: A Prospective, Multi-Center, Randomized, Open-Label, Parallel Group, Superiority Clinical Trial
Brief Title: Transanal Tube Drainage in Endoscopic Submucosal Dissection of the Colorectal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Zhongshan Hospital Endoscopy center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2016-11
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Tumor
Keywords: ESD;Transanal Tube Drainage;Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transanal Tube Drainage (Experimental): patients with transanal tube drainage after ESD
  Interventions: Device: Transanal Tube Drainage
- Without Transanal Tube Drainage (No Intervention): patients without transanal tube drainage after ESD

INTERVENTIONS:
Device: Transanal Tube Drainage — Using transanal tube drainage after colorectal ESD
  Arms: Transanal Tube Drainage

SUMMARY:
We design the clincal trial to investigate the efficacy of transanal tube drainage in colorectal ESD.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a technique for endoscopic tissue resection that enables endoscopists to control the depth and direction of diathermic knife incisions.Recently, the number of reports in which ESD has been successfully used to treat colorectal tumors has increased. But the complatios with colorectal ESD were higher than esophagus and stomach ESD.We design the clincal trial to investigate the efficacy of transanal tube drainage in colorectal ESD.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopy proven colorectal polyp>2cm, LST>3cm, SMTs<2cm Suitable for ESD No other organic disease of colorectal Removing a single lesion one time Informed consent

Exclusion Criteria:

* Complicated other colorectal diseases, such as,Crohn's disease Familial adenomatous polyposis With previous colorectal surgery Pregnancy or lactation Absolute contraindications to general anesthesia or prolonged pneumoperitoneum (ASA class > III) ESD conversion to laparotomy Patients cannot receive ESD Patients and/or family members can not understand and accept this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30 days post operatively
  bleeding, perforation,coagulation syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Center, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No